CLINICAL TRIAL: NCT05458960
Title: Evaluating the Impact of Basic Needs Assessment and Support to Improve Colposcopy Show Rate: The BASICS Trial
Brief Title: Impact of Basic Needs Assessment and Support to Improve Colposcopy Show Rate
Acronym: BASICS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Staffing issues
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202205183; 1R03TR004017-01A1 (NIH)
Record Dates: First submitted 2022-07-08; First posted 2022-07-14 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer
Keywords: Colposcopy; Cervical cancer prevention; Adherence to follow-up; Unmet social needs; Distress
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Social needs navigator program (Experimental): Participants will be paired with a community health worker who will provide tailored support to address unmet social needs. The number and frequency of calls will be limited only by participants' needs, interest, and willingness to interact. The type of contact could include phone calls, or home/community visits. The community health worker will: (1) identify and assess patients' unmet social needs; (2) jointly generate solutions; (3) help prioritize among multiple needs; (4) identify community resources that could help resolve the problem(s); (5) determine eligibility for services; (6) help patients access available resources by scheduling appointments and providing appointment reminders; (7) prepare patients to interact with service agencies and/or act as an advocate; (8) provide support such as arranging transportation; (9) oversee follow-up problem-solving actions; and (10) review progress made towards resolving unmet social needs and adapt solutions.
  Interventions: Behavioral: Social needs navigator program
- Arm 2: Enhanced usual care (Active Comparator): Participants will receive verbal referral to a federally funded, free, 24-hr assistance hotline, United Way 2-1-1, which connects callers with community services to help address unmet social needs.
  Interventions: Behavioral: Enhanced usual care
- Arm 3: Clinic provider (No Intervention): 4 WUSM colposcopy providers, 4 staff members, and 1 community health worker will be surveyed to assess potential for dissemination.

INTERVENTIONS:
Behavioral: Social needs navigator program — 4 months of assistance tailored to the needs of the participant
  Arms: Arm 1: Social needs navigator program
Behavioral: Enhanced usual care — Referral to United Way 2-1-1
  Arms: Arm 2: Enhanced usual care

SUMMARY:
The investigators will perform a randomized controlled trial in which 72 eligible patients (low-income, uninsured, or on Medicaid) who are referred for colposcopy at Washington University School of Medicine, are enrolled and then screened for unmet social needs and distress. The participants will then be randomized 1:1 into either receive the social needs navigator program (n=36) or enhanced usual care (n=36).

ELIGIBILITY:
Inclusion Criteria:

* Abnormal cervical cancer screen
* Missed appointment at BJH colposcopy clinic and need to reschedule
* Age 21 years or older
* Able to provide verbal consent
* Diagnosis of an abnormal cervical screen confirmed by cytology or pathology

Exclusion Criteria:

* Individual without a cervix
* Known diagnosis or history of cancer
* Unable to consent

Ages: 21 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Adherence to colposcopy visit as measured as number of participants who complete colposcopy visit | 6 weeks after enrollment

SECONDARY OUTCOMES:
Total number of unmet basic needs | 4 months after enrollment
  -Unmet basic needs include food security, housing, personal safety, neighborhood safety, sufficient money for necessities, childcare (if applicable), and transportation. A questionnaire will be given to participants to identify the number of unmet basic needs the participant has.
Change in general distress scores as measured by the NCCN Distress Thermometer and Problem List | Enrollment and 4 months after enrollment
  Participants will be asked to rate the amount of distress (scale of 0 to 10, 10=extreme distress) that they have experienced in the past week and the amount of distress (scale of 0 to 10) that they attribute to their abnormal cervical cancer screen. The NCCN distress problem list is a 40-item list categorized into five themes-practical, family, emotional, spiritual, and physical problems¬-and leaves room for patients to describe "other".
Intent to use intervention over time | Completion of study enrollment (estimated to be 18 months)
  -Providers are asked after completion of enrollment to indicate on a scale of 1=not committed to 10=fully committed of how committed they are to use the intervention in their clinic.
Patients' satisfaction with intervention | Completion of study enrollment (estimated to be 18 months)
  -The interview guide has two questions that relate to patient satisfaction related to the intervention. 1) Was the [community health worker or 2-1-1 operator] helpful to you? 2) Would you recommend [the community healthworker/2-1-1] to a family member or friend?
Providers' satisfaction with intervention | Completion of study enrollment (estimated to be 18 months)
  -Providers are asked after completion of enrollment to indicate their satisfaction with the intervention. They are given 12 statements about the satisfaction of the intervention and are asked to circle responses of 1=completely disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, or 5=completely agree. The higher the score the more satisfied the provider is with the intervention.
Resources needed to sustain intervention | Completion of study enrollment (estimated to be 18 months)
  -Validated questionnaire that will be administered to providers, staff, and community health workers: Self-administered 15-minute online survey that will be completed at the end of the study enrollment period. The survey will ask about specific implementation outcomes using the Acceptability Intervention Measure, the Intervention Appropriateness Measure, and the Feasibility of Intervention Measure.
Likelihood that intervention will become built into usual care | Completion of study enrollment (estimated to be 18 months)
  -Providers are asked after completion of enrollment to indicate the likelihood that the intervention can be built into usual care in their clinic. The responses are either likely, very likely, neutral, unlikely, very unlikely, or unsure.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay M Kuroki, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu